CLINICAL TRIAL: NCT02278003
Title: A Pilot Study to Assess the Amnesic Properties of Propofol in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-006
Record Dates: First submitted 2014-10-24; First posted 2014-10-29 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2017-06

CONDITIONS: Pediatric Pateints; Amnesic Properties of Propofol
Keywords: Amnesic; Propofol; 12-006
MeSH Terms: interventions — Propofol

ARMS (2):
- children going under sedation with propofol (Experimental): Children who will undergo sedation as part of their clinical management and give them a memory encoding task during propofol infusion to measure the effects of sedation. The mere task of naming a picture will encode that picture into memory. When the anesthesia has worn off (at approximately 1 hour later), children will be given a memory recognition task to measure the amnesic effects of propofol.
  measure the amnesic effects of propofol.
  Interventions: Other: memory test; Drug: Propofol
- children not going under sedation (Active Comparator): A control group of children of similar age and undergoing similar minor therapeutic procedures will be recruited to perform memory.
  Interventions: Other: memory test

INTERVENTIONS:
Other: memory test
Drug: Propofol
  Arms: children going under sedation with propofol

SUMMARY:
The goal of this study is to extend findings of propofol's effects on memory, as measured in volunteer research studies, to a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be between 4 and 14 yrs of age and be undergoing a therapeutic or diagnostic procedure with or without sedation
* The patient must be able to comprehend and perform the task (naming pictures)
* The patient must have a minimum weight of 8 kg

Exclusion Criteria:

* Allergy to propofol (for those patients requiring sedation)
* Procedure of short duration (< 15 min)
* Pregnancy
* Recent use (within 5 half-lives) of centrally acting medications that could affect concentration (e.g. diphenhydramine)

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Kelhoffer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Veselis R, Kelhoffer E, Mehta M, Root JC, Robinson F, Mason KP. Propofol sedation in children: sleep trumps amnesia. Sleep Med. 2016 Nov-Dec;27-28:115-120. doi: 10.1016/j.sleep.2016.10.002. Epub 2016 Oct 22. PMID 27938911
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Children Going Under Sedation With Propofol: Children who will undergo sedation as part of their clinical management and give them a memory encoding task during propofol infusion to measure the effects of sedation. The mere task of naming a picture will encode that picture into memory. When the anesthesia has worn off (at approximately 1 hour later), children will be given a memory recognition task to measure the amnesic effects of propofol.
  measure the amnesic effects of propofol.
  memory test
  Propofol
- Children Not Going Under Sedation: A control group of children of similar age and undergoing similar minor therapeutic procedures will be recruited to perform memory.
  memory test
Period: Overall Study
Arm/Group | Children Going Under Sedation With Propofol | Children Not Going Under Sedation
Started | 49 | 20
Completed | 30 | 20
Not Completed | 19 | 0
Not completed — Withdrawal by Subject | 11 | 0
Not completed — Not Treated | 1 | 0
Not completed — Recognition task improperly completed | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Children Going Under Sedation With Propofol | Children Not Going Under Sedation | Total
Number analyzed (Participants) | 30 | 20 | 50
Age, Continuous [Mean (Full Range); unit: years] | 6.2 [4.2 to 11.0] | 8.8 [4.4 to 12.6] | 7.2 [4.2 to 12.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 16 | 9 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 26 | 18 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 26 | 18 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 20 | 50

OUTCOME MEASURES:

1. Primary Outcome: Sedation Threshold
Description: During the 10-minute infusion of propofol, children will be presented with pictures at 5-second intervals and asked to name the picture. They will be asked to name each picture (e.g., cat, tree, pencil, etc.). A valid response is naming of the picture within 5 seconds, either correctly or incorrectly.The important response measure is whether the child is awake enough to perform the naming task.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Children Going Under Sedation With Propofol | Children Not Going Under Sedation
Number analyzed (Participants) | 30 | 20
Participants
  Memory Lost w/in 2 minutes of sedation | 29 | NA — This objective is only applicable to participants undergoing sedation.
  No memory loss w/in 2 minutes of sedation | 1 | 0

2. Secondary Outcome: Memory Threshold
Description: At the presentation of each picture, the child will be asked whether or not he/she remembers having seen it previously. Each response will be coded as correct (true positives and true negatives) or incorrect (false positives and false negatives).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Hit rate
Arm/Group | Children Going Under Sedation With Propofol | Children Not Going Under Sedation
Number analyzed (Participants) | 30 | 20
Hit rate | 0.71 (0.16) | 0.93 (0.06)

ADVERSE EVENTS:
Time Frame: AE data was collected on the day of treatment. There is no follow-up period.
Arm/Group | Children Going Under Sedation With Propofol | Children Not Going Under Sedation
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/20
Other Adverse Events (participants affected / at risk) | 0/30 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT02278003/Prot_SAP_000.pdf